CLINICAL TRIAL: NCT07229586
Title: A Phase IB/II Clinical Study of the Safety, Tolerability and Efficacy of SHR-7367 in Combination With Anti-tumor Agents in Subjects With Solid Tumors
Brief Title: A Study of SHR-7367 With Anti-tumor Agents in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-4642-205-01
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Paclitaxel; Injections; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-7367 + SHR-1316 Group (Experimental): SHR-7367 combined with SHR-1316.
  Interventions: Drug: SHR-7367 Injection; Drug: SHR-1316 Injection
- SHR-7367 + SHR-1316 + AG Group (Experimental): SHR-7367 combined with SHR-1316 and AG.
  Interventions: Drug: SHR-7367 Injection; Drug: SHR-1316 Injection; Drug: Paclitaxel for Injection; Drug: Gemcitabine Hydrochloride for Injection
- SHR-7367 + AG Group (Experimental): SHR-7367 combined with AG.
  Interventions: Drug: SHR-7367 Injection; Drug: Paclitaxel for Injection; Drug: Gemcitabine Hydrochloride for Injection

INTERVENTIONS:
Drug: SHR-7367 Injection — SHR-7367 injection.
Drug: SHR-1316 Injection — SHR-1316 injection.
  Arms: SHR-7367 + SHR-1316 + AG Group; SHR-7367 + SHR-1316 Group
Drug: Paclitaxel for Injection — Paclitaxel for injection (Albumin Bound).
  Arms: SHR-7367 + AG Group; SHR-7367 + SHR-1316 + AG Group
Drug: Gemcitabine Hydrochloride for Injection — Gemcitabine Hydrochloride for injection.
  Arms: SHR-7367 + AG Group; SHR-7367 + SHR-1316 + AG Group

SUMMARY:
This study aims to evaluate the safety and preliminary efficacy of SHR-7367 in combination with antineoplastic agents in subjects with advanced solid tumors, and to determine the maximum tolerated dose (MTD) and the recommended Phase II dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide a written informed consent.
2. Age 18-75 years old (inclusive) at the time of signing the informed consent form.
3. ECOG performance status 0-1.
4. Life expectancy is not less than 12 weeks.
5. At least one measurable lesion per RECIST v1.1.
6. Adequate organ and marrow function as defined by the protocol.

Exclusion Criteria:

1. Presence of uncontrollable psychiatric illness and other conditions such as known alcoholism, drug or substance abuse, criminal detention, etc., that affect the completion of the study procedures.
2. Known hypersensitivity to any component of SHR-7367; History of severe allergic reactions to other monoclonal antibodies/fusion protein drugs; Known history of severe hypersensitivity to antineoplastic agents in combination.
3. Subjects who are participating in other clinical studies or whose first dose is less than 4 weeks from the end of the previous clinical study (last dose).
4. Surgery or chemotherapy within 4 weeks of the first dose of study treatment.
5. Active HBV/HCV/HIV infection.
6. Untreated and/or uncontrolled brain metastases.
7. Any other condition that, in the judgment of the investigator, may increase the risk of participating in the study, interfere with the results of the study, or be unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Stage 1 (IB Period): Dose-limiting toxicity (DLT). | Up to 28 days.
Stage 1 (IB Period): Adverse events (AEs). | About 1 year.
Stage 1 (IB Period): Serious adverse events (SAEs). | About 1 year.
Phase II: Investigator-assessed objective response rate (ORR). | Assessed every 6 weeks, about 1 year.

SECONDARY OUTCOMES:
Investigator-assessed objective response rate (ORR). | Assessed every 6 weeks, about 1 year.
  Complete response + Partial response (CR+PR) based on RECIST v1.1.
Disease control rate (DCR). | Assessed every 6 weeks, about 1 year.
  Complete response + Partial response + Stable disease (CR+PR+SD) based on RECIST v1.1.
Duration of response (DoR). | Assessed every 6 weeks, about 1 year.
  Time from documentation of tumor response to disease progression assessed among patients who had an objective response.
Progression Free Survival (PFS). | Assessed every 6 weeks, about 1 year.
  Time from C1D1 to the first assessment of disease progression or death, whichever is earlier.
Incidence and severity of Adverse events (AEs). | Assessed approximately once every 1 month, about 1 year.
  Time from C1D1 to the first assessment of disease progression or death, whichever is earlier.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided